CLINICAL TRIAL: NCT05579184
Title: Phase 2 Study of Repeat-dose [177Lu]Ludotadipep Treatment for Metastatic Castration-resistant Prostate Cancer
Brief Title: [Lu-177]Ludotadipep in Castration-resistant Prostate Cancer(CRPC): Investigation of Drug and Application_2
Acronym: LUCIDA_2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: FutureChem (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FC705-2
Record Dates: First submitted 2022-10-06; First posted 2022-10-13 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer, mCRPC
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [177Lu]Ludotadipep 100 mCi (Experimental): 100 mCi of [177Lu] ludotadipep shall be administered to the subject repeatedly up to 6 times at intervals of 8 weeks (±2 weeks).
  Interventions: Drug: [177Lu]Ludotadipep

INTERVENTIONS:
Drug: [177Lu]Ludotadipep — Patients will receive 100 mCi of [177Lu]Ludotadipep every 8 [±1] weeks (up to 6 times)
  * Test article code/name: [177Lu]Ludotadipep
  * Administration route: intravenous injection
  * Total dose strength: 4 to 6 x 3.7 GBq
  * Dosage form: solution for injection

SUMMARY:
100 mCi of [177Lu]Ludotadipep, the dose determined in the phase 1 clinical trial (FC705-1), was administered repeatedly up to 6 times at intervals of 8 weeks (±2 weeks) to patients with metastatic castration resistant prostate cancer (mCRPC) in order to assess the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male over the age of 19 as of the date of written consent
2. Adenocarcinoma confirmed by histopathology or cytology
3. Those who have been confirmed with at least two metastases in the soft tissue lesions or bone lesions based on the PCWG3 modified RECIST v1.1 criterion for prostate adenocarcinoma, or those who experience pain due to radiologically apparent disease progression
4. Those with castration resistance with a blood testosterone level of 50 ng/dL or less at the time of screening and those who meet one or more of the criteria below

   * Prostate cancer patients with resistance against imaging-based progression of metastatic castration even after at least 4 weeks of imaging-based progression of standard medical treatment using one or more second-generation hormonal agents (e.g., enzalutamide, abiraterone) are administered in combination with standard taxene-based chemotherapy (e.g., docetaxel).

     * In cases where the patient is judged unsuitable by the investigator for the standard medical treatment specified above

       * In cases where the patient himself/herself refuses the standard medical treatment specified above
5. Those that exhibit lesions of 4 or higher PSMA reporting and data system (P-RADS) in the [18F] PSMA PET/CT imaging at the time of screening
6. Those that exhibit higher or wider uptake of the lesion in [18F] PSMA PET/CT imaging than [18F] FDG PET taken at the time of screening as judged by the investigator
7. Those who exhibit an ECOG performance score of level 2 or less at the time of screening and with an expected survival period of at least 6 months
8. Subjects having active sexual activities with a fertile female spouse must satisfy the following:

   * If the spouse is a fertile woman (including pregnant and lactating women), the subject must consent to maintain abstinence or to use double contraception* from the time of screening and throughout the entire clinical trial period and at least 6 months after the administration of the last investigational drug.
   * Sperm of the subject must not be donated during the entire clinical trial period from the time of screening and for at least 6 months after the administration of the last investigational drug.

     * Double contraception: If applicable to at least two of the following: the use of condoms, non-hormonal intrauterine device, diaphragm, cervical cap, if it has been more than 3 months since the male spouse had a vasectomy (at the time of initial screening visit), or the spouse is medically diagnosed with infertility
9. Those who have fully understood the purpose, details, and characteristics of the investigational drug from the investigator before enrolling in the clinical trial and signed the informed consent form in person or by guardian or legal representative

Exclusion Criteria:

1. Those who are judged to have abnormalities in bone marrow, liver, or kidney function as they are in accordance with the results of laboratory tests that satisfy at least one of the following criteria at the time of screening:

   * If ANC is below 1.5 x 109/L

     * If Hemoglobin is below 9.0 g/dL

       * If the platelet count is below 100 x 109/L

         * If total bilirubin exceeds 1.5 times the normal value,

           * If serum albumin is below 2.5 g/dL

             * If the glomerular filtration rate (eGFR) is below 50 mL/min
2. Those with one or more of the following diseases at the time of screening

   * Those who correspond to Classification III-IV under the New York Heart Association (NYHA) classification of patients with severe heart failure

     * Patients with uncontrolled hypertension (SBP > 160 mm Hg or DBP > 90 mm Hg)

       * Patients with uncontrolled diabetes (HbA1c > 7.0% or fasting blood sugar > 160 mg/dL)
3. Those with a history of prostate cancer or solid cancer other than radical metastasis limited to bone or soft tissue with basis on prostate cancer or blood cancer including lymphoma within 3 years from the time of screening (However, non-melanoma skin cancer, superficial bladder cancer, thyroid cancer, and intraepithelial carcinoma (carcinoma in situ) that do not require continued treatment as they are treated appropriately and remain disease-free within 2 years from the time of screening)
4. Those who have received radiopharmaceutical treatment or radiotherapy for the target lesion of metastatic prostatic carcinoma within 12 weeks from the time of screening
5. Those with active infection of HIV, HBV, HCV, or VDRL at the time of screening, or those with other uncontrolled active infectious diseases with proteinuria of > 1.0 in protein under the urine protein vs. creatinine ratio
6. Those suffering from one or more disease of the following: Immunosuppressive status (including nephrectomy, hematopoietic stem cell transplantation) and autoimmune disease patients (including severe myasthenia, Hashimoto thyroiditis, rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosus, scleroderma) at the time of screening
7. Those who had participated in a therapeutic clinical trial within 30 days of screening and had been administered or applied with other investigational products or investigational devices.
8. Those with potential hypersensitivity reaction to this investigational product [177Lu] ludotadipep
9. Those with an anamnesis of clinically significant mental illness, alcohol abuse, etc.
10. Those who are judged unsuitable by the investigator to participate in this clinical trial for other miscellaneous reasons or who are judged incompatible with the administration requirements

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients aged 19 years or older
Enrollment: 20 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prostate-Specific Antigen Response Rate (PSA-RR) | up to 48 weeks (Response Rate from Baseline to EOT(End of Treatment))
  Defined as the proportion of participants with a PSA reduction of ≥ 50% from baseline

SECONDARY OUTCOMES:
Prostate-Specific Antigen Response Rate (PSA-RR) | Between 4 and 6 weeks after treatment
  The prostate-specific antigen response rate (PSA-RR) is assessed after the administration of [177Lu]Ludotadipep
Changes in the Standardized Uptake Values (SUV) of [18F]PSMA PET/CT | up to 48 weeks (up to 6 doses at 8-weekly intervals [± 1 week], with 6 week follow-up after each dose (Screening up to 28 days)
  The tumor response is assessed by comparing the changes in the Standardized Uptake Values (SUV) of [18F]PSMA PET/CT after administration of [177Lu]Ludotadipep compared to pre-administration
Objective Response Rate (ORR) | up to 48 weeks (up to 6 doses at 8-weekly intervals [± 1 week], with 6 week follow-up after each dose (Screening up to 28 days)
  The objective response rate (ORR) is assessed after administration of [177Lu]Ludotadipep
The Best Objective Response Rate (BORR) | up to 48 weeks (up to 6 doses at 8-weekly intervals [± 1 week], with 6 week follow-up after each dose (Screening up to 28 days)
  The best objective response rate (BORR) is assessed after administration of [177Lu]Ludotadipep
Progression-Free Survival (PFS) | up to 48 weeks (up to 6 doses at 8-weekly intervals [± 1 week], with 6 week follow-up after each dose (Screening up to 28 days)
  The imaging-based progression-free survival (PFS) is assessed after administration of [177Lu]Ludotadipep
Objective Response Rate (ORR) | up to 48 weeks (up to 6 doses at 8-weekly intervals [± 1 week], with 6 week follow-up after each dose (Screening up to 28 days)
  The objective response rate (ORR) is assessed while using PCWG3 modified RECIST V1.1 after administration of [177Lu]Ludotadipep
Pain response rate | up to 48 weeks (up to 6 doses at 8-weekly intervals [± 1 week], with 6 week follow-up after each dose (Screening up to 28 days)
  ≥2 point reduction in Present Pain Intensity Scale (PPI) score from baseline with no increase in analgesic score; and/or ≥50% decrease in analgesic score with no increase in PPI using the McGill Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ji Youl Lee, Ph.D, Principal Investigator — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea, Seoul, St, Mary's Hospital, 222, Banpo-daero, Seocho-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No